CLINICAL TRIAL: NCT00429845
Title: Effect of Nutritional Intervention on the Lipid Profile of HIV-Positive Patients Who Start on Highly Active Antiretroviral Therapy: a Randomized Trial
Brief Title: Effect of Nutritional Intervention on the Lipid Profile of HIV-Positive Patients Who Start HAART: a Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HCPA2004-012
Record Dates: First submitted 2007-01-30; First posted 2007-02-01 (Estimated); Last update posted 2007-02-01 (Estimated); Status verified 2007-01

CONDITIONS: HIV Infections
Keywords: HIV; HAART; Nutrition; Dyslipidemia
MeSH Terms: conditions — HIV Infections; Dyslipidemias

INTERVENTIONS:
Behavioral: Nutritional

SUMMARY:
Highly active antiretroviral therapy (HAART) in HIV-positive patients is associated with the development of dyslipidemia, a risk factor for cardiovascular events. The objective of this study was to evaluate the effect of dietary intervention in individuals who start HAART.

DETAILED DESCRIPTION:
Adult patients prescribed to HAART that met the exclusion criteria were consecutively enrolled in a randomized trial:

* control (receiving general guidelines on dietary education)
* intervention (receiving general guidelines on dietary education and nutritional follow-up every 3 months)

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive individuals naive to HAART, with clinical indication to start therapy

Exclusion Criteria:

* Diabetes Mellitus
* Pregnancy
* Active opportunistic disease
* Any mental deficiency
* Use of lipid profile influencing drugs
* Use of illicit drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2004-03; Study Completion 2007-02

PRIMARY OUTCOMES:
Total cholesterol and of triglycerides levels

SECONDARY OUTCOMES:
HDL-cholesterol, LDL-cholesterol, weight, waist to hip ratio

CONTACTS AND LOCATIONS:
Overall Officials: Jorge P Ribeiro, MD, ScD, Principal Investigator — Associate Professor and Chief of Non-invasive Cardiology
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Lazzaretti RK, Kuhmmer R, Sprinz E, Polanczyk CA, Ribeiro JP. Dietary intervention prevents dyslipidemia associated with highly active antiretroviral therapy in human immunodeficiency virus type 1-infected individuals: a randomized trial. J Am Coll Cardiol. 2012 Mar 13;59(11):979-88. doi: 10.1016/j.jacc.2011.11.038. PMID 22402068